CLINICAL TRIAL: NCT00754962
Title: A Single Dose, 2-Period, 2-way Crossover Bioequivalency Study of Protriptyline Tablets 10 mg Under Fasted Conditions
Brief Title: Bioequivalency Study of Protriptyline 10 mg Tablets Under Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director - Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PROT-T10-PVFS-1
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Protriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: protriptyline — 10 mg tablet
  Other Names: Vivactil

SUMMARY:
The objective of this study was to prove the bioequivalence of Protriptyline 10 mg tablets under fasted conditions

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to Protriptyline or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2006-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | baseline, 2-period, 28 day washout

CONTACTS AND LOCATIONS:
Overall Officials: Benno G Roesch, MD, Principal Investigator — Advanced Biomedical Research
Locations (1):
- Advanced Biomedical Research, Hackensack, New Jersey, United States